CLINICAL TRIAL: NCT00370994
Title: A Randomized, Prospective, Double-blind Controlled Evaluation of the Effectiveness of Percutaneous Lumbar Epidural Adhesiolysis and Hypertonic Saline Neurolysis
Brief Title: Effectiveness of Percutaneous Lumbar Epidural Adhesiolysis and Neurolysis on Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pain Management Center of Paducah (Other)
Responsible Party: Principal Investigator, Laxmaiah Manchikanti, MD, Medical Director, Pain Management Center of Paducah
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: protocol 11
Record Dates: First submitted 2006-08-30; First posted 2006-09-01 (Estimated); Results first posted 2015-11-23 (Estimated); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Low Back Pain
Keywords: post-lumbar surgery syndrome; percutaneous lumbar epidural adhesiolysis; hypertonic saline neurolysis
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Caudal epidural injection (Active Comparator): Caudal epidural with placement of catheter in sacral canal with injection of 5 mL of 2% preservative-free lidocaine, followed by 6 mL of 0.9% sodium chloride solution and 6 mg of non-particulate Betamethasone and 1 mL of sodium chloride solution
  Interventions: Procedure: Caudal epidural injection
- Percutaneous adhesiolysis (Active Comparator): Pecutaneous adhesiolysis and targeted placement of Racz catheter with injection of 5 mL of 2% preservative-free lidocaine, followed by 6 mL of 10% sodium chloride solution and 6 mg of non-particulate Betamethasone and 1 mL of sodium chloride solution
  Interventions: Procedure: Percutaneous adhesiolysis

INTERVENTIONS:
Procedure: Caudal epidural injection — Caudal epidural injection with catheterization
  Arms: Caudal epidural injection
Procedure: Percutaneous adhesiolysis — Percutaneous adhesiolysis with hypertonic saline neurolysis
  Arms: Percutaneous adhesiolysis

SUMMARY:
Clinically significant improvements in the percutaneous adhesiolysis patients with hypertonic neurolysis compared to those patients randomized to the control group who did not receive adhesiolysis and hypertonic saline neurolysis. Improvement will be assessed in relation to the clinical outcome measures of pain and function.

Improvements among patients with adhesiolysis and hypertonic saline neurolysis and compare to control group.

Compare adverse event profile in both groups

DETAILED DESCRIPTION:
Patients with chronic low back pain and lower extremity pain secondary to spinal stenosis or post lumbar laminectomy syndrome, non responsive to conservative therapy with physical therapy or chiropractic and medical therapy and fluoroscopically directed epidural steroid injections.

Single-center, prospective, controlled, double blind, randomized study. If non-responsive or at patient's request, the patient may be unblinded anytime after 3 months, and will be offered adhesiolysis and hypertonic saline neurolysis if the patient was in the control group. All patients will be unblinded at 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age
* History of chronic, function limiting low back pain of at least 6 months in duration
* Able to give voluntary, written informed consent
* Able to understand investigational procedures and willing to return for follow-ups
* No recent surgical procedures within last 3 months

Exclusion Criteria:

* Large contained or sequestered herniation
* Cauda Equina symptoms and/or compressive radiculopathy
* Narcotic use of no greater than 100mg/day Hydrocodone, 60mg Methadone, or 100mg Morphine
* Uncontrolled major depression or psychiatric disorder
* Uncontrolled or acute medical illness
* Chronic sever conditions that could interfere with outcome assessments
* Women who are pregnant or lactating
* Subjects who have participated in a clinical study with an investigational product within 30 days of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2006-01; Primary Completion 2009-12 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laxmaiah Manchikanti, MD, Principal Investigator — Ambulatory Surgery Center
Locations (1):
- Ambulatory Surgery Center, Paducah, Kentucky, United States

REFERENCES:
- [Result] Manchikanti L, Singh V, Cash KA, Pampati V. Assessment of effectiveness of percutaneous adhesiolysis and caudal epidural injections in managing post lumbar surgery syndrome: 2-year follow-up of a randomized, controlled trial. J Pain Res. 2012;5:597-608. doi: 10.2147/JPR.S38999. Epub 2012 Dec 20. PMID 23293536
- [Derived] Manchikanti L, Singh V, Cash KA, Pampati V, Datta S. A comparative effectiveness evaluation of percutaneous adhesiolysis and epidural steroid injections in managing lumbar post surgery syndrome: a randomized, equivalence controlled trial. Pain Physician. 2009 Nov-Dec;12(6):E355-68. PMID 19935992
- [Derived] Manchikanti L, Cash KA, McManus CD, Pampati V, Singh V, Benyamin R. The preliminary results of a comparative effectiveness evaluation of adhesiolysis and caudal epidural injections in managing chronic low back pain secondary to spinal stenosis: a randomized, equivalence controlled trial. Pain Physician. 2009 Nov-Dec;12(6):E341-54. PMID 19935991
- See also: Assessment of effectiveness of percutaneous adhesiolysis and caudal epidural injections in managing post lumbar surgery syndrome: 2-year follow-up of a randomized, controlled trial. — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC3533727/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: An interventional pain management practice, a specialty referral center, a private practice setting in the United States
Groups:
- Pecutaneous Adhesiolysis: Pecutaneous adhesiolysis and targeted placement of Racz catheter with injection of 5 mL of 2% preservative-free lidocaine, followed by 6 mL of 10% sodium chloride solution and 6 mg of non-particulate Betamethasone and 1 mL of sodium chloride solution
Period: Overall Study
Arm/Group | Caudal Epidural Injection | Pecutaneous Adhesiolysis
Started | 60 (Sample size was 200, due to the difficulties of recruiting we changed to 120) | 60
Completed | 60 | 60
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Caudal Epidural Injection | Pecutaneous Adhesiolysis | Total
Number analyzed (Participants) | 60 | 60 | 120
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 44 | 48 | 92
  >=65 years | 16 | 12 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 52 (13.9) | 52 (12.5) | 52 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 35 | 70
  Male | 25 | 25 | 50
Region of Enrollment [Number; unit: participants]
  United States | 60 | 60 | 120

OUTCOME MEASURES:

1. Primary Outcome: Numeric Pain Rating Score
Description: Numeric rating scale represented 0 with no pain and 10 with the worst pain imaginable
Time Frame: 3, 6, 12, 18 and 24 months post treatment.
Population: Sample size is calculated based on reduction of NRS. A 25% clinical difference change of 1.15.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Control Group: caudal epidural injections since no adhesiolysis was performed and there was no injection of 10% sodium chloride solution.
- Intervention Group: adhesiolysis and targeted placement of Racz catheter with injection of 5 mL of 2% preservative-free lidocaine, followed by 6 mL of 10% sodium chloride solution and 6 mg of non-particulate Betamethasone and 1 mL of sodium chloride solution
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 60 | 60
units on a scale
  Baseline | 7.9 (0.8) | 8.1 (0.8)
  3 months | 4.9 (1.6) | 3.4 (0.8)
  6 months | 5.8 (1.5) | 3.7 (1.1)
  12 months | 6.1 (1.4) | 4.0 (1.2)
  18 months | 6.1 (1.4) | 3.6 (1.2)
  24 months | 6.2 (1.4) | 3.6 (1.2)
Statistical Analysis 1: Comparison: Control Group vs Intervention Group; Test type: Superiority or Other; p < 0.001, Repeated measures ANOVA. — Comparisons were made between groups and within the group between baseline and different time points

2. Secondary Outcome: Functional Status
Description: Oswestry Disability Index (ODI) - ODI score is ranged from 0 to 50. Total score is converted in to percent disability. ODI Scoring: 0% to 20% (minimal disability), 21%-40% (moderate disability), 41%-60% (severe disability), 61%-80% (crippled) and 81%-100 These patients are either bed-bound or exaggerating their symptoms.
Time Frame: 3, 6, 12, 18 and 24 months post treatment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 60 | 60
units on a scale
  Baseline | 28.6 (4.1) | 31.2 (4.1)
  3 months | 20.2 (6.6) | 15.2 (4.1)
  6 months | 22.3 (6.1) | 15.2 (5.2)
  12 months | 23.3 (5.8) | 15.8 (5.6)
  18 months | 23.3 (5.7) | 14.6 (4.6)
  24 months | 23.2 (6.7) | 13.9 (5.1)
Statistical Analysis 1: Comparison: Control Group vs Intervention Group; Test type: Superiority or Other; p = 0.001, Repeated measures of ANOVA — There were significant differences in Oswestry Disability Index between both groups

ADVERSE EVENTS:
Arm/Group | Caudal Epidural Injection | Pecutaneous Adhesiolysis
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/60
Other Adverse Events (participants affected / at risk) | 0/60 | 0/60

LIMITATIONS AND CAVEATS:
The results of this study are limited by potentially inadequate double blinding, by the lack of a placebo group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes